CLINICAL TRIAL: NCT04915209
Title: Integrated Parkinson Care Networks: Addressing Complex Care in Parkinson Disease in Contemporary Society
Brief Title: Integrated Parkinson Care Networks : Care in Parkinson Disease
Acronym: ICARE-PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/19/0489
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
Keywords: healthcare
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Narrative interviews
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Narrative interviews (Other): Narratives are stories that are based on the unfolding of events or actions from the perspective of a patient's life experience. Patients and care partners tell their stories of illness and how they live with illness over time . The researcher could focus on the care priorities, the support needed, the information needed and the challenges faced. The narrative interview will be used to get an overview of the patient's trajectory.
  Interventions: Other: Narrative interviews

INTERVENTIONS:
Other: Narrative interviews — During the workshop, the participants will collectively create a common representation of the patient journey and co-design the envisioning care delivery model that support both social care and medical care.

SUMMARY:
The researchers wish to determine what are patients/care partners priorities in terms of care delivery based at home/community and define the envisioning care delivery model that support both social care and medical care from the perspective of people living with Parkinson.

DETAILED DESCRIPTION:
The researchers wish to determine what are patients/care partners priorities in terms of care delivery based at home/community and define the envisioning care delivery model that support both social care and medical care from the perspective of people living with Parkinson.

Narrative interviews and workshops are conducted to obtain information on:

1. Everyday life, living with PD (perception and consequences of PD in everyday life)
2. Care delivery priorities from the perspective of PwPs & Care Partners
3. Factors influencing care delivery (facilitators & barriers)
4. Needs and expectations about social care and medical care
5. Role playing by eHealth technologies in a care delivery model based at home/community

Narratives are stories that are based on the unfolding of events or actions from the perspective of a patient's life experience. Patients and care partners tell their stories of illness and how they live with illness over time. They are encouraged to share their personal stories of living with PD, using health services, community resources.

The researcher could focus on the care priorities, the support needed, the information needed and the challenges faced. The narrative interview will be used to get an overview of the patient's trajectory.

During the workshop, the participants will collectively create a common representation of the patient journey and co-design the envisioning care delivery model that support both social care and medical care.

A patient journey map gives a common picture of the process and the way patients experience their care delivery. Understanding the patients' experiences of their journey is essential in order to co-design the future care delivery model based at home/community.

Journey map proposes a visual representation of the relationship between patients and the healthcare services. They also help to visually externalize patient experience by placing them at the heart of the modelling process. The journey map is an effective tool that reduces the complexity of health services to a comprehensible representation.

At the end of the workshop, patients' needs and care priorities will be discussed considering the different phases of the patient journey, and the participants will be encouraged to envisioning the future care delivery model based at home/community.

ELIGIBILITY:
Inclusion Criteria:

* Major patients, over 18 and under 65 years of age, Diagnosed at different stages of Parkinson's disease (recent, intermediate, advanced) Understands and speaks French to be able to answer questionnaires and interviews Affiliated to a social security scheme Patient who did not oppose participation in the study. Where possible, we will vary the profiles of people: socio-demography, gender, age, etc.

Exclusion Criteria:

* Patient and/or participant objecting to the research Pregnant and/or nursing women Persons under justice, guardianship or curatorship In-patient or intensive care patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-22 (Estimated); Primary Completion 2021-12-22 (Estimated); Study Completion 2022-12-22 (Estimated)

PRIMARY OUTCOMES:
Narrative interviews | 1 day
  Identify the expectations and priorities of people living with Parkinson's disease for medical-social benefits.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Rascol, MD PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France